CLINICAL TRIAL: NCT04596059
Title: A Retrospective and Comparative Study on the Journey of Children With Cow´s Milk Protein Allergy in Mexico: Current Practice in Allergy Management in Mexican Children Aged ≤24 Months
Brief Title: The Journey of Children With Cow's Milk Protein Allergy in Mexico.
Acronym: Friso02
Status: Completed | Type: Observational
Sponsor: FrieslandCampina (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: CEI00320171130/07/052020
Record Dates: First submitted 2020-10-02; First posted 2020-10-22 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frisolac Gold Intensive HA — Regular medical care
  Other Names: Frisolac Gold PEP AC

SUMMARY:
To gain insights on the application, use and effectiveness of Frisolac Gold Intensive HA and Frisolac Gold PEP AC with reference to improvement of CMPA symptoms and to determine the methodology used by Mexican Health Care Professionals (HCPs) in the clinical practice (i.e. diagnosis and dietary management) of CMPA in Mexican children (≤24 months) diagnosed with or suspected of CMPA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with electronic/physical medical records that contain sufficient data to answer the primary question (i.e. data on growth and dermatological symptoms (based on the SCORAD score) at diagnosis and follow up data of at least 2 months or successful completion of therapy according to the PI (whichever comes first).
* Subjects ≤24 months of age at the moment of suspected or diagnosed CMPA with records available between January 2016 to September 2020.
* Subjects prescribed with Frisolac Gold Intensive HA and/or Frisolac Gold PEP AC for the dietary management of their CMPA symptoms.

Exclusion Criteria:

* Subjects using other formula products/breast milk alongside Frisolac Gold Intensive HA or Frisolac Gold PEP AC during the time of their participation in the study.
* Premature children, or children with low birth-weight (weight at birth <2.5 kg).
* Subjects diagnosed with a metabolic condition that impacts development and growth.
* Subjects diagnosed with a congenital condition and/or with prior or current disease that in the opinion of the PI could potentially interfere with their participation in the study.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Mexican children (≤24 months) diagnosed with or suspected of CMPA.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Growth | Can be 2 weeks up to 2 months
  * the proportion of subjects with weight gain compared to the previous visit (%)
  * the proportion of subjects with height gain compared to the previous visit (%)
  * the proportion of subjects with both weight and height gain compared to the previous visit (%)
Dermatological symptoms (SCORAD score) | Can be 2 weeks up to 2 months
  The proportion of subjects with an 1-point improvement in their SCORAD intensity category in between 2 visits (%)

SECONDARY OUTCOMES:
Type of symptoms | Can be 2 weeks up to 2 months
  Type of symptoms (e.g. crying, regurgitation, stool consistency, respiratory, enteropathies and colitis) (based on clinical diagnosis)
Number of symptoms | Can be 2 weeks up to 2 months
  Number of symptoms (e.g. crying, regurgitation, stool consistency, respiratory, enteropathies and colitis) (based on clinical diagnosis)
Severity of symptoms | Can be 2 weeks up to 2 months
  Severity of symptoms on first and second visit (based on clinical diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa E Huerta Hernandez, MD, Principal Investigator — Clínica de Alergia Pediátrica, México; Benjamin Zepeda Ortega, MD, Principal Investigator — Clinica San Antonio, Mexico; Marlene Ruiz Castillo, MD, Principal Investigator — Hospital del Niño DIF Hildago, Mexico; Consultorio de Pediatría Pachuca, Mexico
Locations (4):
- Mexico (4):
  - Clinica San Antonio, Mexico City
  - Clínica de Alergia Pediátrica, Pachuca
  - Consultorio de Pediatria, Pachuca
  - Hospital del Niño DIF, Pachuca

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estrada Reyes E, Zepeda Ortega B, Ten Haaf D, Kudla U, Muhardi L, Hofman DL, Hageman JHJ, Huerta Hernandez RE. Symptom's resolution and growth outcome of children with cow's milk protein allergy consuming two hydrolyzed formulas: A retrospective study in Mexico. Front Allergy. 2023 Jan 30;4:1073430. doi: 10.3389/falgy.2023.1073430. eCollection 2023. PMID 36793546